CLINICAL TRIAL: NCT07345481
Title: The Principle of Stimulus Equivalence Learning and Its Neuropsychological Correlates in Adults With Acquired Brain Injury (ABI).
Brief Title: Stimulus Equivalence Learning in Acquired Brain Injury.
Status: Recruiting | Type: Observational
Sponsor: Klimmendaal Revalidatiespecialisten (Network)
Collaborators: Donders Centre for Cognitive Neuroimaging (Other)
Responsible Party: Sponsor
Other Study IDs: KNP23PROJ2
Record Dates: First submitted 2025-12-10; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Acquired Brain Injury (Including Stroke)
Keywords: acquired brain injury; implicit memory
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy controls
- acquired brain injury

SUMMARY:
Stimulus Equivalence Learning (SEL) is a form of learning in which stimuli (such as words, pictures, or sounds) become linked to one another in memory, even though this specific connection has not been directly taught. In a typical SEL task, two relations are taught explicitly (A→B and A→C), and the untrained relation (B→C) is then tested. This indirect relation is not intentionally or consciously learned and is considered a form of implicit learning. The principle of stimulus equivalence learning is still rarely applied in cognitive rehabilitation after acquired brain injury (ABI), with the exception of a few small (N=1) treatment studies that have shown positive effects. However, it remains unclear to what extent ABI may affect the ability to acquire stimulus equivalence.

ELIGIBILITY:
Inclusion Criteria:

ABI patients (>3 months post-injury), including stroke, traumatic brain injury, brain tumor, encephalitis, and out-of-hospital cardiac arrest (OHCA).

Exclusion Criteria:

Neurodegenerative disorders Severe psychiatric disorders (including suicidality) Insufficient command of the Dutch language Severe cognitive impairments, aphasia, or visual or hearing problems that make test administration impossible

An additional exclusion criterion for controls was any medical condition that could lead to cognitive impairment beyond normal aging, including stroke, TBI, brain tumor, or other forms of brain injury.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ABI patients (>3 months post-injury), including stroke, traumatic brain injury, brain tumor, encephalitis, and out-of-hospital cardiac arrest (OHCA).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Modified Rutgers Equivalence Learning Task (mRAET) | Day 1
  The original RAET is an experimental paradigm in which faces have to be paired with colored fish. For the current study, this task has been adapted into a more ecologically valid version focused on medication intake, in which relationships are learned between the shape of a pill, the function of the pill, the time of intake, and the (fictional) brand name.

SECONDARY OUTCOMES:
Location Learning Test (LLT) | Day 1
  The LLT is a test that can be used to measure episodic spatial memory for object locations. Normalized scores for immediate and delayed spatial memory are computed (percentiles 0-100).
Wechsler Adult Intelligence Scale IV-NL digit span (WAIS-IV-NL DS) | Day 1
  The digit span is a measure of verbal working memory. Normalized standard scores can be computed (range 0-19, mean: 10, standard deviation: 3).
Everyday memory questionnaire-revised (EMQ-R) | Day 1
  This is a 13-item scale of the everyday memory functioning.
Trial Making Test | Day 1
  The Trail Making Test (TMT) is a neuropsychological test that measures processing speed, visual attention, and task switching.
Stroop | Day 1
  The Stroop Test is a cognitive task that measures selective attention, processing speed, and the ability to inhibit automatic responses. Participants are shown color words printed in incongruent ink colors (e.g., the word "red" printed in blue ink) and must name the ink color rather than read the word. The interference effect-slower or less accurate responses-reflects challenges in cognitive control and response inhibition.
Rey Auditory Verbal Learning Test (RAVLT) | Day 1
  The Rey Auditory Verbal Learning Test, RAVLT) is a verbal learning and memory task in which a list of 15 unrelated words is read aloud over several trials. The participant is asked to recall as many words as possible after each trial, and later again after a delay. The test assesses immediate recall, learning ability, retention, and recognition memory.
Serial Reaction Time Task (SRTT) | Day 1
  Participants respond to the location of a black circle that appears in one of four screen positions by pressing the corresponding response key as quickly and accurately as possible. After 12 practice trials, the task consists of 8 blocks of 60 trials.
  Blocks 1-6 contain a fixed repeating sequence of locations (not disclosed to participants). Block 7 contains a different sequence, followed by a return to the original sequence in Block 8. After the task, participants complete questions assessing explicit awareness of the sequence.
  Implicit learning is indicated by faster reaction times in Blocks 6 and 8 (repeated sequence) compared to Block 7 (irregular sequence).

CONTACTS AND LOCATIONS:
Locations (1):
- Klimmendaal Revalidatiespecialisten, Arnhem, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided